CLINICAL TRIAL: NCT06586112
Title: A Multicenter, Randomized, Double-Blind, Placebo and Active Comparator Controlled Phase 3 Study to Evaluate the Efficacy and Safety of ESK-001 in Patients With Moderate to Severe Plaque Psoriasis (ONWARD1)
Brief Title: A Study to Evaluate the Efficacy and Safety of ESK-001 in Patients With Moderate to Severe Plaque Psoriasis
Acronym: ONWARD1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESK-001-016
Record Dates: First submitted 2024-08-14; First posted 2024-09-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ESK-001 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- Placebo (Placebo Comparator): Matching oral placebo
  Interventions: Drug: Placebo
- Apremilast (Active Comparator): Apremilast administered as an oral capsule
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: ESK-001 — ESK-001
  Arms: ESK-001
Drug: Apremilast — Apremilast
  Arms: Apremilast
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if ESK-001 works to treat moderate to severe plaque psoriasis. The main questions it aims to answer are:

* Does ESK-001 reduce the severity of people's psoriasis?
* How safe is ESK-001 in people with moderate to severe plaque psoriasis?

The study includes 2 comparators: a placebo control (a 'dummy' tablet that does not contain the medicine ESK-001 but looks just like it) and an active control (apremilast, which is a medicine approved to treat psoriasis).

People taking part in this study must be men or women aged at least 18 years and have had plaque psoriasis for at least 6 months, currently moderate to severe.

Participants will:

* take drug every day for 24 weeks.
* visit the clinic for checkups and tests.
* fill out questionnaires about their psoriasis, itch severity, and change in quality of life.
* be assessed for health issues and side effects, physical examinations, vital signs, heart electrical activity measurements, and psychological health.
* provide blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age ≥18 years
2. Diagnosis of plaque psoriasis for ≥6 months
3. Plaques covering ≥10% of BSA
4. PASI ≥12
5. sPGA ≥3
6. Women of childbearing potential (WOCBP) and males who are sexually active with WOCBP must agree to adhere to highly effective methods of contraception

Exclusion Criteria:

1. Nonplaque psoriasis or other inflammatory skin conditions
2. immune-mediated conditions commonly associated with psoriasis (eg inflammatory bowel disease). Participants with psoriatic arthritis may participate
3. Pregnant, lactating, or planning to get pregnant during the study
4. Use of drugs prior to Study Day 1 that treat or may affect psoriasis:

   * Topical within 2 weeks
   * Phototherapy or any systemic treatments within 4 weeks
   * Any biologic agent targeted to IL-12 or IL-23 within 6 months, oral IL-12 or IL-23 or TNFα inhibitor within 2 months, or IL-17 within 4 months
   * Systemic immunosuppressants or immunomodulatory drugs within 4 weeks
   * Modulators of B cells within 6 months, or T cells within 3 months
   * JAK inhibitors or TYK2 inhibitors within 4 weeks
   * PDE4 inhibitor within 2 months
   * Any investigational agent, within 30 days or 5 half-lives or is currently enrolled in an investigational study
5. Lack of clinical response to a TYK2, IL-12, or IL-23 targeted psoriasis treatment
6. Participants with QTcF >450 msec (males) or >470 msec (females) at Screening
7. Unstable cardiovascular disease, defined as a recent clinical deterioration or a cardiac hospitalization within the last 3 months
8. Evidence of recent or recurrent herpes zoster or herpes simplex viral infection
9. Evidence of active infection or positive test result for hepatitis B, hepatitis C, HIV or TB
10. History of serious bacterial, fungal, or viral infections that led to hospitalization, or any recent serious infection requiring antibiotic treatment
11. Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status
12. Lab abnormalities indicating significant renal, hepatic or bone marrow dysfunction
13. History of any immune-mediated or inflammatory medical condition for which participants requires current systemic corticosteroids

    * Stable doses of inhaled corticosteroids for treatment of asthma are allowed
14. Known current malignancy or current evaluation for a potential malignancy or history of malignancy within the past 5 years prior to screening, except for adequately treated basal cell or squamous cell skin carcinoma or carcinoma in situ of the cervix
15. Live vaccines within 4 weeks prior to Study Day 1
16. Participant has planned surgery during the study period
17. Any acute or chronic illness/condition or evidence of an unstable clinical condition that, in the opinion of the Investigator, will substantially increase the risk to the participant if he or she participates in the study
18. History of mental illness within the last 5 years, unless receiving a fixed regimen of psychiatric medications for at least 6 months before screening or has not required or been prescribed any psychiatric medication within 12 months before screening
19. Evidence of severe depressive symptoms or active suicidal ideation or behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether ESK-001 reduces the severity of psoriasis by 75% (using the PASI) or by at least 2 points (using sPGA score) compared to placebo | 16 weeks
  Proportion of participants achieving ≥75% reduction in PASI score. Proportion of participants achieving a score of 0 or 1 on sPGA.

SECONDARY OUTCOMES:
To compare the Psoriasis Area and Severity Index (PASI-90 and PASI-100) between ESK-001 and placebo or apremilast | 24 weeks
  Proportion of participants achieving of ≥90% or 100% reduction in PASI
To compare the Psoriasis Area and Severity Index (PASI-75) between ESK-001 and apremilast | 24 weeks
  Proportion of participants achieving of ≥75% reduction in PASI
To compare the Static Physician's Global Assessment (sPGA-0/1) between ESK-001 and apremilast | 24 weeks
  Proportion of participants achieving a score of 0 or 1 on sPGA
To compare the affected body surface area (%BSA) between ESK-001 and placebo or apremilast | 24 weeks
  Change from baseline in %BSA
To compare the scalp specific Physician's Global Assessment (ssPGA) between ESK-001 and placebo or apremilast. | 24 weeks
  Proportion of participants achieving a score of 0 or 1 on ssPGA
To compare the Psoriasis Symptoms and Signs Diary (PSSD) between ESK-001 and placebo or apremilast | 24 weeks
  Proportion of participants achieving a score of 0
To compare the Dermatology Life Quality Index (DLQI) between ESK-001 and placebo or apremilast | 24 weeks
  Proportion of participants achieving a score of 0 or 1
To compare the Pruritus numeric rating scale (NRS) between ESK-001 and placebo | 24 weeks
  Change from baseline in Pruritus NRS
Proportion of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 24 weeks
  Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)
To characterize the pharmacokinetics of ESK-001 | 24 weeks
  Maximum [Cmax] and minimum [Cmin] plasma concentration

CONTACTS AND LOCATIONS:
Locations (158):
- United States (55):
  - Alliance Dermatology, Phoenix, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Northwest Arkansas Clinical Trials Center (NWACTC), PLLC, Rogers, Arkansas
  - Exalt Clinical Research, Chula Vista, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Marvel Clinical Research, LLC, Huntington Beach, California
  - Sunwise Clinical Research, LLC, Lafayette, California
  - Wallace Medical Group Inc, Los Angeles, California
  - Northridge Clinical Trials - Elite Clinical Network, Northridge, California
  - Pasadena Clinical Trials, Pasadena, California
  - Therapeutics Clinical Research, San Diego, California
  - Unison Clinical Trials/ Shahram Jacobs MD, Sherman Oaks, California
  - Olive View - UCLA Education & Research Institute, Sylmar, California
  - California Dermatology Institute - Thousand Oaks, Thousand Oaks, California
  - Clearlyderm Dermatology - West Boca Raton, Boca Raton, Florida
  - Driven Clinical Research, Coral Gables, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Glick Skin Institute - Margate, Margate, Florida
  - San Marcus Research Clinic, Inc - Miami, Miami Lakes, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - Oceanic Research Group, North Miami Beach, Florida
  - LENUS Research, Sweetwater, Florida
  - Caban Skin Institute, Tampa, Florida
  - ForCare Medical Center, Tampa, Florida
  - Skin Care Physicians of Georgia - Warner Robins, Macon, Georgia
  - MetroMed Clinical Trials, Chicago, Illinois
  - Arlington Dermatology, Rolling Meadows, Illinois
  - NorthShore Medical Group - Dermatology - Skokie, Skokie, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group, Columbus, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - Equity Medical - Bowling Green, Bowling Green, Kentucky
  - Velocity Clinical Research at The Dermatology Clinic, Baton Rouge, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - MetroBoston Clinical Partners, Brighton, Massachusetts
  - Cleaver Dermatology, Kirksville, Missouri
  - OptiSkin, New York, New York
  - The Ohio State University Wexner Medical Center (OSUWMC) - OSU Dermatology East - Columbus, Gahanna, Ohio
  - Dermatologists of Southwestern Ohio, LLC, Mason, Ohio
  - Unity Clinical Research (UCR), Oklahoma City, Oklahoma
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Paddington Testing Company Inc., Philadelphia, Pennsylvania
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Discover Dermatology, LLC d/b/a Goodlettsville Dermatology Research, Goodlettsville, Tennessee
  - Discover Dermatology, LLC d/b/a Cumberland Skin Center for Clinical Research under Objective Health, Hermitage, Tennessee
  - UT Health Houston Department of Dermatology, Bellaire, Texas
  - Studies in Dermatology, LLC, Cypress, Texas
  - Reveal Research Institute, Frisco, Texas
  - Center for Clinical Studies - Texas Medical Center, Houston, Texas
  - Austin Institute for Clinical Research - Houston, Houston, Texas
  - University of Utah Health Care - Midvalley Health Center, Murray, Utah
  - Frontier Dermatology, Mill Creek, Washington
- Australia (5):
  - Premier Specialists, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - North Eastern Health Specialists (NEHS), Campbelltown, South Australia
  - Skin Health Institute Inc., Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment Dr Tota Venkova, Gabrovo, Gabrovo
  - Clineca, Stara Zagora, Stara Zagora
  - Medikal Center Kordis, Pleven
  - Skin and Venereal Diseases Center EOOD, Sofia
  - Diagnostic Consultative Center Aleksandrovska EOOD, Sofia
- Canada (15):
  - Rejuvenation Medical Group Edmonton Downtown, Edmonton, Alberta
  - Enverus Medical Research, Surrey, British Columbia
  - Dermatrials Research Inc., Hamilton, Ontario
  - Centricity Research, London, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - Institute of Cosmetic & Laser Surgery, Oakville, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - North York Research Inc., Toronto, Ontario
  - Canadian Dermatology Centre, Toronto, Ontario
  - Dermatology on Bloor, Toronto, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - "Centre de Recherche Dermatologique du Quebec Metropolitain Inc.", Québec, Quebec
  - Dermatologie Sima Inc., Verdun, Quebec
- Czechia (16):
  - Fakultni nemocnice Plzen Dermatovenerologicka klinika, Pilsen, Bory
  - Pratia Brno s.r.o., Brno, Moravia
  - Dermskin, s.r.o., Olomouc, Moravia
  - Kozni ambulance Kutna Hora, s.r.o., Kutná Hora
  - DERMAMEDICA, s.r.o., Náchod
  - Nemocnice Nový Jičín, A.S., Nový Jičín
  - CCR Ostrava, s.r.o., Ostrava
  - Vesalion sro, Ostrava
  - Pratia Pardubice a.s., Pardubice
  - Clintrial s.r.o., Prague
  - Fakultni Nemocnice Kralovske Vinohrady FNKV Dermatovenerologicka Klinika, Prague
  - Sanatorium Profesora Arenbergera, Prague
  - Pratia Prague, s.r.o., Prague
  - Praglandia, Prague
  - Dermatologicka ambulance - Svitavy, Svitavy
  - MUDr Radka Neumannova, Svitavy
- Germany (11):
  - Eberhard Karls Universitaet Tuebingen Universitaets Hautklinik Tuebingen, Tübingen, Baden-Wurttemberg
  - Hautarztpraxis Dr. Mihaescu, Augsburg, Bavaria
  - Hautarztpraxis Mahlow, Mahlow, Brandenburg
  - Universitatsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Hautarztpraxis an der Hase, Bramsche, Lower Saxony
  - Siteworks, Lohne, Lower Saxony
  - Klinikum Bielefeld, Bielefeld, North Rhine-Westphalia
  - Pro Derma, Dülmen, North Rhine-Westphalia
  - Intramedis CSS, Remscheid, North Rhine-Westphalia
  - Universitatsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
- Japan (19):
  - Fukuoka University Hospital, Fukuoka, Fukuoka-shi
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-Ku
  - Saruwatari Dermatology Clinic, Kagoshima, Kagoshima-Shi
  - Kanto Rosai Hospital, Kanagawa, Kawasaki-shi
  - Nagoya City University Hospital, Aichi, Nagoya-shi
  - Okayama University Hospital, Okayama, Okayama-shi
  - Osaka Metropolitan University Hospital, Osaka, Osaka-shi
  - Nippon Life Hospital, Osaka, Osaka-Shi
  - National Hospital Organization Sagamihara National Hospital, Kanagawa, Sagamihara
  - Dermatology and Ophthalmology Kume Clinic, Osaka, Saka-Shi
  - Hokkaido University Hospital, Hokkaido, Sapporo-shi
  - Kindai University Hospital, Osaka, Sayama-Shi
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-Ku
  - Osaka University Hospital, Osaka, Suita-shi
  - Medical Corporation Jitai kai Tachikawa Dermatology Clinic, Tokyo, Tachikawa-shi
  - Mie University Hospital, Mie, Tsu-shi
  - Yamaguchi University Hospital, Yamaguchi, Ube-shi
  - Yokohama City University Hospital, Kanagawa, Yokohama-shi
- Poland (21):
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczny Ośrodek Alergologiczno-Internistyczny "ALL-MED", Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Synexus Wroclaw, Wroclaw, Lower Silesian Voivodeship
  - WroMedica, Wroclaw, Lower Silesian Voivodeship
  - Diamond Clinic, Krakow, Malopolska
  - MICS Medical Center Warsaw, Warsaw, Masovian Voivodeship
  - FutureMeds Warszawa Centrum, Warsaw, Masovian Voivodeship
  - High Med Przychodnia Specjalistyczna, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park, Warsaw, Masovian Voivodeship
  - RoyalDerm, Warsaw, Mazowiecke
  - ClinicMed Daniluk, Nowak Spolka Komandytowa, Bialystok, Podlaskie Voivodeship
  - AES Gdansk, Gdansk, Pomeranian Voivodeship
  - Derm Art Institute, Gdynia, Pomeranian Voivodeship
  - Centrum Medyczne Synexus Gdynia, Gdynia, Pomeranian Voivodeship
  - Centrum Medyczne Angelius Provita (Angelius Provita Medical Centre), Katowice, Silesian Voivodeship
  - Laser Clinic, Szczecin, West Pomeranian Voivodeship
  - Centrum Badań Klinicznych PI House Sp. Z O.O., Gdansk
  - Pratia Małopolskie Centrum Medyczne (MCM) Kraków, Krakow
  - Rheuma Medicus, Warsaw
  - Centrum Medyczne Synexus Warszawa, Warsaw
  - Velocity Clinical Research, Skierniewice, Skierniewice, Łódź Voivodeship
- Portugal (3):
  - Hospital da Senhora da Oliveira, Guimarães, Braga District
  - Hospital CUF Descobertas, Lisbon, Lisbon District
  - Unidade Local de Saude Santo Antonio Hospital de Santo Antonio, Porto, Porto District
- South Korea (8):
  - Chosun Universtiy Hospital, Gwangju, Dong-gu
  - Konkuk University Medical Center, Seoul, Gwangjin-gu
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Kyung Hee University Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
The Sponsor Alumis Inc. is a clinical-stage biopharmaceutical company that has not yet adopted an Individual Participant Data (IPD) sharing plan.